CLINICAL TRIAL: NCT05809310
Title: The Effects of Branch Pulmonary Artery Stenting in d-TGA, ToF and TA: a Randomized Control Trial
Brief Title: Effects Branch PA Stenting d-TGA, ToF and TA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Heart Foundation (Other); Hartekind (Unknown); Erasmus Medical Center (Other); Leiden University Medical Center (Other); Amsterdam University Medical Centers (UMC), Location Academic Medical Center (AMC) (Other)
Responsible Party: Principal Investigator, Hans Breur, Dr., UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL81160
Record Dates: First submitted 2023-03-15; First posted 2023-04-12 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Transposition of Great Vessels; Tetralogy of Fallot; Truncus Arteriosus; Pulmonary Artery Stenosis Supravalvular Congenital; Stent Stenosis; Right Ventricular Dysfunction; Congenital Heart Disease
Keywords: Exercise capacity
MeSH Terms: conditions — Transposition of Great Vessels; Tetralogy of Fallot; Truncus Arteriosus, Persistent; Ventricular Dysfunction, Right; Heart Defects, Congenital | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Percutaneous intervention for PA stenosis
  Interventions: Procedure: Percutaneous intervention (stent) for PA stenosis
- Control group (No Intervention): Conservative management (percutaneous intervention for PA stenosis 6 months postponed)

INTERVENTIONS:
Procedure: Percutaneous intervention (stent) for PA stenosis — Percutaneous intervention (stent placement) in one or both of the branch pulmonary arteries
  Arms: Interventional group

SUMMARY:
The goal of this randomized controlled trial is to identify the effects of percutaneous interventions for branch PA stenosis on exercise capacity in patients with d-TGA, ToF and TA.

The main question[s] it aims to answer are:

The primary study objective is to identify the effects of percutaneous interventions for branch PA stenosis on exercise capacity in patients with d-TGA, ToF and TA. The secondary objectives are 1) to assess the effects of percutaneous interventions for branch PA stenosis on RV function and 2) to define early markers for RV function and adaptation to improve timing of these interventions.

Participants will undergo the same series of examinations at baseline and approximately 6 months follow-up (within 6 week time-range) as part of standard care: conventional transthoracic echocardiogram (TTE), cardiopulmonary exercise testing (CPET) and conventional Cardiac Magnetic Resonance (CMR) including a low dose dobutamine stress MRI to assess RV functional reserve. The low dose dobutamine stress MRI will be performed in the interventional group from the UMC Utrecht/WKZ and Erasmus MC because the LUMC and AUMC do not have a suitable infrastructure for the low dose dobutamine stress MRI and this cannot be achieved throughout the duration of this study. The baseline CMR in the interventional group will be performed as close as possible prior to the intervention but maximal 4 weeks prior to the intervention. In addition, the intervention group will undergo standard RV pressure measurements during the intervention. Quality of life (QoL) questionnaires will be obtained at baseline and 2 weeks post intervention (intervention group) or a similar time range in the control group, which is based on experts opinion. TTE, CPET and conventional CMR will be performed within 2-4 years follow-up to assess the long-term effects of percutaneous PA interventions.

Researchers will compare the difference in VO2 max (% predicted) between the interventional group (TGA, ToF or TA patients with a class II indication for a PA intervention who will undergo a percutaneous intervention for a PA stenosis) and the control group (TGA, ToF or TA patients with a class II indication for a PA intervention who will undergo conservative management)

DETAILED DESCRIPTION:
Rationale: Postoperative survival of patients with dextro transposition of the great arteries (d-TGA), Tetralogy of Fallot (ToF) and Truncus Arteriosus (TA) has increased over the last decades due to advances in operative techniques and perioperative care. Despite postoperative survival has increased, morbidity of these patients increases during long-term follow-up with a high need for reinterventions. Right ventricular outflow tract (RVOT) obstructions are the most common indication for a reintervention and percutaneous branch pulmonary artery (PA) interventions account for a significant number of these reinterventions. However, the effects of percutaneous branch PA interventions on exercise capacity, RV function and RV adaptation of patients with d-TGA, ToF and TA remains largely unknown. In addition, there is no consensus about the optimal timing for percutaneous interventions for branch PA stenosis in international guidelines.

Objective: The primary study objective is to identify the effects of percutaneous interventions for branch PA stenosis on exercise capacity in patients with d-TGA, ToF and TA. The secondary objectives are 1) to assess the effects of percutaneous interventions for branch PA stenosis on RV function and 2) to define early markers for RV function and adaptation to improve timing of these interventions.

Study design: This is a multicenter randomized controlled trial. Patients will be included from the following Dutch interventional centers for congenital heart disease: UMC Utrecht/WKZ (sponsor), LUMC/AUMC and Erasmus MC. During this trial there will be two groups: 1. a group of patients with d-TGA, ToF and TA who will undergo a percutaneous intervention for a branch PA stenosis according to standard care (intervention group) and 2. a group of patients with d-TGA, ToF and TA with a similar degree of pulmonary stenosis as group 1 (class IIa indication) who will undergo conservative management for a branch PA stenosis according to standard care (control group). If necessary, the control group will be able to undergo a percutaneous intervention for branch PA stenosis after the examinations at approximately 6 months follow-up, or sooner in case of symptoms. Patients from both groups will undergo the same series of examinations at baseline and approximately 6 months follow-up (within 6 week time-range) as part of standard care: conventional transthoracic echocardiogram (TTE), cardiopulmonary exercise testing (CPET) and conventional Cardiac Magnetic Resonance (CMR) including a low dose dobutamine stress MRI to assess RV functional reserve. The low dose dobutamine stress MRI will be performed in the interventional group from the UMC Utrecht/WKZ and Erasmus MC because the LUMC and AUMC do not have a suitable infrastructure for the low dose dobutamine stress MRI and this cannot be achieved throughout the duration of this study. The baseline CMR in the interventional group will be performed as close as possible prior to the intervention but maximal 4 weeks prior to the intervention. In addition, the intervention group will undergo standard RV pressure measurements during the intervention. Quality of life (QoL) questionnaires will be obtained at baseline and 2 weeks post intervention (intervention group) or a similar time range in the control group, which is based on experts opinion. TTE, CPET and conventional CMR will be performed within 2-4 years follow-up to assess the long-term effects of percutaneous PA interventions.

Study population: d-TGA post ASO, ToF or TA patients ≥8 years old will be included if they have a class IIa indication for a percutaneous intervention for branch PA stenosis according to the international guidelines. Patients will be excluded if they contraindications for one of the examinations.

Main study parameters/endpoints: the difference in VO2 max (% predicted) as parameter for exercise capacity between the interventional and control group.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Patients with d-TGA post ASO, ToF or TA
* ≥8 years

Exclusion Criteria:

One or more of the following inclusion criteria:

* All class IIa indications for a branch PA intervention:
* Persistent decreased RV function (based on gold standard CMR)

  * <18 years RVEF ≤55% (28)
  * ≥18 years RVEF<50% (29)
* Progressive tricuspid regurgitation (TR) (≥moderate)
* Isolated bifurcation stenosis:

  * Significant unilateral stenosis (≥50%)
  * Borderline bilateral PA stenosis (40-70%)
* Unbalanced perfusion (≤35/65%)
* RV/LV pressure ratio > 2/3 based on echocardiography
* Reduced lung perfusion or decreased objective exercise capacity (based of gold standard VO2 max during CPET)

  * <18 years VO2 peak <35 mL∙kg-1∙min-1 (boys) VO2 peak <30 mL∙kg-1∙min-1 (girls) (30)
  * ≥18 years VO2 peak <27 mL∙kg-1∙min-1 (men) VO2 peak <19 mL∙kg-1∙min-1 (women) (31)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline VO2max as percentage of predicted at 6 months as indication of exercise capacity | change between baseline and 6 months follow-up
  using cardiopulmonary exercise test on a treadmill

SECONDARY OUTCOMES:
Technical success using invasive right ventricular and pulmonary artery pressures and gradients | after the intervention, an average of 1 month after baseline
  Technical success of the intervention using invasive right ventricular and pulmonary artery pressures and gradients
Peak workload (W) | at baseline, 6 months follow-up and 2-4 years follow-up
  using cardiopulmonary exercise test on a treadmill
Peak workload (% predicted) | at baseline, 6 months follow-up and 2-4 years follow-up
  using cardiopulmonary exercise test on a treadmill
O2 pulse (ml) | at baseline, 6 months follow-up and 2-4 years follow-up
  using cardiopulmonary exercise test on a treadmill
O2 pulse (% predicted) | at baseline, 6 months follow-up and 2-4 years follow-up
  using cardiopulmonary exercise test on a treadmill
VE/VCO2 slope | at baseline, 6 months follow-up and 2-4 years follow-up
  using cardiopulmonary exercise test on a treadmill
Right ventricular ejection fraction (%) | at baseline, 6 months follow-up and 2-4 years follow-up
  using CMR
RV strain (%) | at baseline, 6 months follow-up and 2-4 years follow-up
  using speckle tracking echocardiography and CMR feature tracking
RV fractional area change (%) | at baseline, 6 months follow-up and 2-4 years follow-up
  using echocardiography
RV pressure (mmHg) | at baseline, 6 months follow-up and 2-4 years follow-up
  using echocardiography (TI gradient)
RV end-systolic elastance | before and after the intervention, an average of 1 month after baseline
  using pressure-volume analysis
RV end systolic volume (ml and ml/m2) | at baseline, 6 months follow-up and 2-4 years follow-up
  using CMR
RV end diastolic volume (ml and ml/m2) | at baseline, 6 months follow-up and 2-4 years follow-up
  using CMR
RV functional reserve | at baseline and 6 months follow-up in the interventional group from UMC Utrecht and Erasmus MC
  RVEF dobutamine - RVEF rest using a low dose dobutamine stress MRI
RV mass (g and g/m2) | at baseline, 6 months follow-up and 2-4 years follow-up
  using CMR
Right ventricular pulmonary arterial (RV-PA) coupling | before and after the intervention, an average of 1 month after baseline
  using pressure-volume analysis
Lung perfusion (%) | at baseline, 6 months follow-up and 2-4 years follow-up
  using CMR
Quality of Life (QoL) in 4 domains: health and related activities, emotional, social and school/work | at baseline and 2 weeks follow-up
  using PedsQL questionnaire

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Amsterdam University Medical Center location AMC, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam
  - UMC Utrecht/WKZ, Utrecht

IPD SHARING:
Plan to Share IPD: No
We will publish the results in peer-reviewed journals and present them at meetings and conferences. As the data is privacy-sensitive, the database will not be publically available. A request for a collaboration can be made via DataverseNL.

REFERENCES:
- [Derived] Joosen RS, Voskuil M, Krasemann TB, Blom NA, Krings GJ, Breur JMPJ; Outreach consortium. The effects of percutaneous branch pulmonary artery interventions in biventricular congenital heart disease: study protocol for a randomized controlled Dutch multicenter interventional trial. Trials. 2024 Sep 3;25(1):581. doi: 10.1186/s13063-024-08436-8. PMID 39227910